CLINICAL TRIAL: NCT04576026
Title: Effect of Exogenous Ketone Supplementation on Cognitive Function During Exercise After Induced Mental Fatigue
Brief Title: Exogenous Ketone Supplementation and Cognitive Function During Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Professor, Western University, Canada
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 116711
Record Dates: First submitted 2020-09-29; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Ketonemia; Mental Fatigue; Ketosis
Keywords: Ketone supplements; Cognitive function; Exercise
MeSH Terms: conditions — Ketosis; Mental Fatigue; Motor Activity | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: This will be a double blind repeated measures cross over study. There will be two treatments involved: Ketone esters supplements and iso-caloric carbohydrates (placebo). Participants will complete the protocol twice and the treatment order will be systematically rotated to avoid any order effect. Design of the study is composed of a mental fatiguing task, followed by a 45 minute simulated soccer game (second half). Cognitive function will be assessed during the 45 minutes of exercise. All participants will perform the protocol in a fed state (4 h after consumption of their last meal)
Who Masked: Participant, Investigator
Masking Description: Participants and investigators will be blinded as an individual not involved in the project will assemble and distribute the treatment (drinks) according to a coding system that is kept confidential until the study is completed. Participants will complete the protocol twice and the treatment order will be systematically rotated to avoid any order effect. taste and texture of treatments will be matched and will be distribute in opaque bottles to keep participant blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone esters (Experimental): Ketone esters will be given to mentally fatigued individuals, prior to a 45 minute simulated soccer game in which cognitive function will be assessed.
  Interventions: Behavioral: mental fatiguing task; Behavioral: 45 - minute simulated soccer game; Behavioral: cognitive function
- Placebo (Active Comparator): Iso-caloric carbohydrate drink will be given to mentally fatigued individuals, prior to a 45 minute simulated soccer game in which cognitive function will be assessed.
  Interventions: Behavioral: mental fatiguing task; Behavioral: 45 - minute simulated soccer game; Behavioral: cognitive function

INTERVENTIONS:
Behavioral: mental fatiguing task — a 30-minute computerized Stroop test will be used to induce mental fatigue before exercise intervention
Behavioral: 45 - minute simulated soccer game — an intermittent running protocol using intensities and speeds seen in soccer will be used to simulate the physiological demands of the sport
Behavioral: cognitive function — The Stroop test and a complex reaction time test will be used to assess cognitive function during exercise.

SUMMARY:
15 healthy trained males will volunteer to participate in this study. there will be 2 treatments: Ketone esters supplementation and iso-caloric carbohydrate. The purpose of this study is to evaluate the effect of ketone esters on cognitive function during exercise after induced mental fatigue

DETAILED DESCRIPTION:
mental fatigue is often seen in sports of moderate to long duration. its onset is associated with detriments in cognitive function which leads to poor decision making and detriments in specific sport skills. Ketones can serve as a powerful brain fuel source so they may have the potential to delay/ revert the onset of mental fatigue. in this experiment, we will induce mental fatigue in individuals who will be performing 45 minutes of intermittent exercise right after. During exercise cognitive function will be measured under 2 condition, Ketone supplementation and placebo. The purpose of this study is to see if ketones can play a role in reverting that initial mental fatigue during exercise, compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study you must be a healthy male or female recreationally active individual, 18-35 year old.

Exclusion Criteria:

* You will be excluded from this study if you:
* Are not involved in regular exercise (at least 2x week)
* Have symptoms or take medication for respiratory, cardiovascular, metabolic, neuromuscular disease
* Use any medications with side effects of dizziness, lack of motor control, or slowed reaction time
* Are taking part in another research study
* For women, if you are pregnant or become pregnant during the study.
* Have a history of concussion/head injuries.
* Have an excessive alcohol intake (>2 drinks/day)
* Are consuming a ketogenic diet (for at least 2 weeks)
* Are a smoker
* ** Cannabis use is not a exclusion criteria; however, it must be avoided on experimental days.**

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 30 minutes
  participants will be doing the Stroop test and a complex reaction test during exercise.

SECONDARY OUTCOMES:
Blood Ketones | 45 minutes
  Ketones in blood will be measured using a ketone meter
Blood Glucose | 45 minutes
  blood glucose will be measured using a glucometer
Blood Lactate | 45 minutes
  blood lactate will be measured using a lactate meter

CONTACTS AND LOCATIONS:
Overall Officials: Peter WR Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Laboratory, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No